CLINICAL TRIAL: NCT06165432
Title: Effectiveness of Pre Injection Use of Cryoanesthesia as Compared to Topical Anesthetic Gel in Reducing Pain Perception During Palatal Injections
Brief Title: Pre Injection Use of Cryoanesthesia Versus Topical Anesthetic Gel in Reducing Pain Perception During Palatal Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Siddhartha Rai, Principal investigator, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 556/077/078
Record Dates: First submitted 2023-09-05; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Benzocaine; Ice

STUDY DESIGN:
Intervention Model Description: Cross sectional comparative split mouth study
Who Masked: Outcomes Assessor
Masking Description: Assessment of objective pain using Sound, Eye and Motor scale will be done by a single outcome assessor who will be blinded about the intervention technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug Arm :Topical benzocaine (Active Comparator): since its a split mouth study one half of the hard palate will receive topical benzocaine i.e Group A
  Interventions: Drug: Topical Benzocaine
- Topical ice (Active Comparator): Other half of the palate will receive topical ice i.e Group B
  Interventions: Other: Topical ice

INTERVENTIONS:
Drug: Topical Benzocaine — Benzocaine topical anesthetic gel will be used a pre-injection anesthetic on one half of the palate before giving greater palatine nerve block
  Arms: Drug Arm :Topical benzocaine
Other: Topical ice — For the other half of the palate topical ice would be used before greater palatine nerve block
  Arms: Topical ice

SUMMARY:
The goal of this interventional study is to assess the effectiveness of pre-injection use of topical ice application in decreasing pain perception when administering greater palatine nerve block injections as compared to that of topical 20 % benzocaine anesthetic gel using Visual Analogue Scale (VAS) for subjective pain assessment and Sound, Eye, Motor (SEM) scale for objective pain assessment in adult patients.

The main question it aims to answer are:

1. Does topical cooling reduce pain as effectively as topical benzocaine during greater palatine nerve block injections?
2. Is there any adverse reactions during and after application of topical ice and 20 % benzocaine gel?
3. Is there any difference in patient acceptability to the use of either methods during the administration of greater palatine nerve block.

A split mouth design was used where an anesthetic injection was administered in the left and right posterior palatal area. The same operator administered the injections so as to standardize the flow rate and delivery style. The method of intervention i.e topical ice or topical 20% benzocaine anesthetic gel was randomly allocated to the patient by lottery method. The participants received two palatal injections with an interval of two weeks between the appointments. The subjective pain response of the patients during greater palatine nerve block injection with pre-injection use of topical ice and topical anesthetic gel (20% benzocaine) was recorded using VAS scale. The objective pain response of the patients were recorded by a blinded single observer using SEM scale on the same day of the appointment.

Technique of application of topical ice: A new pack of sterile cotton swabstick that was injected with 0.5ml commercially available bottled water and then freezed the day before the appointment. At the time of intervention the injection site was dried with gauge piece and the frozen cotton swab stick was held by its wooden part and the frozen cotton end was placed on the proposed anesthetic site (palatal mucosa just anterior to the greater palatine foramen) for 1 minute. With the frozen cotton swabstick in place, an injection of 0.5 mL of 2 percent Lidocaine with 1:200,000 epinephrine was administered into the injection site via a 27-gauge short needle.

Technique of application of topical anesthetic gel: After the oral mucosa was dried with a gauze piece, application of 0.2 mL Benzocaine 20% gel was done with a sterile swab stick on the proposed anesthetic site (palatal mucosa just anterior to the greater palatine foramen) for a period of two minutes as shown in figure. With the cotton swabstick in place an injection of 0.5 mL of 2 percent Lidocaine with 1:200,000 epinephrine was administered into the injection site via a 27-gauge short needle.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy patients ASA I and ASA II with intact palatal mucosa on both sides
* Procedures that needs administration of greater palatine nerve block

Exclusion Criteria:

* Hypersensitivity to local anesthetic agent
* Patient who are physically and mentally sub normal
* Presence of palatal mucosal lesions
* Patients on long term neuromodulators for chronic pain
* Patient not consenting to participate in the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
subjective pain perception during greater palatine nerve block injection | Immediatley after the injection
  measured using Visual analogue Scale (VAS) - The Visual Analogue Scale (VAS) consisting of a 100 mm straight line with the endpoints marked to denote extreme limits on the left as 'no pain at all' and on the right as 'pain as bad as it could be' was used to record the pain score . The patient was asked to mark their pain level on the line between the two endpoints after receiving the palatal injection. The distance between 'no pain at all' and the mark defined the subject's pain which was measured in millimeters.
objective pain perception during greater palatine nerve block injection | During the injection procedure
  measured using Sound, Eye and Motor (SEM) scale -The SEM scale was used in the assessment of the relationship between pain and the reactions which the sensation of pain generates in the patient's eyes, bodily movements and verbal expressions of discomfort

SECONDARY OUTCOMES:
Adverse effects | upto 30 minutes after the injection
  Immediate adverse side effects like burning/stinging sensation, local hypersensitivity reaction (urticaria, erythema, itching) and immediate systemic effects (dizziness, drowsiness, palpitations) were assessed; marked as 0: absent and 1: present.
Acceptability regarding the use of either topical ice or topical benzocaine | 5 minutes after application
  The overall patient perception regarding the use of topical ice and topical benzocaine as a preanesthetic agent was assessed using a 5 point Likert scale containing 5 response options that consisted of two extreme sides and a neutral option.
  The five response options were: 1.Very bad, 2 Bad, 3. satisfactory 4. Good and 5. Very Good

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Jaisani, MDS, Study Chair — B.P. Koirala Insititute of Health Sciences
Locations (1):
- B.P Koirala institute of health sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 3 months after publication
Access Criteria: via email

REFERENCES:
- [Background] Hindocha N, Manhem F, Backryd E, Bagesund M. Ice versus lidocaine 5% gel for topical anaesthesia of oral mucosa - a randomized cross-over study. BMC Anesthesiol. 2019 Dec 16;19(1):227. doi: 10.1186/s12871-019-0902-8. PMID 31842771
- [Background] Davoudi A, Rismanchian M, Akhavan A, Nosouhian S, Bajoghli F, Haghighat A, Arbabzadeh F, Samimi P, Fiez A, Shadmehr E, Tabari K, Jahadi S. A brief review on the efficacy of different possible and nonpharmacological techniques in eliminating discomfort of local anesthesia injection during dental procedures. Anesth Essays Res. 2016 Jan-Apr;10(1):13-6. doi: 10.4103/0259-1162.167846. PMID 26957683
- [Background] Kumar M, Chawla R, Goyal M. Topical anesthesia. J Anaesthesiol Clin Pharmacol. 2015 Oct-Dec;31(4):450-6. doi: 10.4103/0970-9185.169049. PMID 26702198
- [Background] Meechan JG. Intra-oral topical anaesthetics: a review. J Dent. 2000 Jan;28(1):3-14. doi: 10.1016/s0300-5712(99)00041-x. PMID 10666956
- [Background] Gondim DGA, Montagner AM, Pita-Neto IC, Bringel RJS, Sandrini FAL, Moreno EFC, de Sousa AM, Correia AB. Comparative Analysis of the Effectiveness of the Topical Administration of Benzocaine and EMLA(R) on Oral Pain and Tactile Sensitivity. Int J Dent. 2018 Feb 7;2018:7916274. doi: 10.1155/2018/7916274. eCollection 2018. PMID 29593794
- [Background] Lee HS. Recent advances in topical anesthesia. J Dent Anesth Pain Med. 2016 Dec;16(4):237-244. doi: 10.17245/jdapm.2016.16.4.237. Epub 2016 Dec 31. PMID 28879311
- [Background] Kosaraju A, Vandewalle KS. A comparison of a refrigerant and a topical anesthetic gel as preinjection anesthetics: a clinical evaluation. J Am Dent Assoc. 2009 Jan;140(1):68-72; quiz 112-3. doi: 10.14219/jada.archive.2009.0020. PMID 19119169
- [Background] Fuzier R, Lapeyre-Mestre M, Mertes PM, Nicolas JF, Benoit Y, Didier A, Albert N, Montastruc JL; French Association of Regional Pharmacovigilance Centers. Immediate- and delayed-type allergic reactions to amide local anesthetics: clinical features and skin testing. Pharmacoepidemiol Drug Saf. 2009 Jul;18(7):595-601. doi: 10.1002/pds.1758. PMID 19402039
- [Background] Lathwal G, Pandit IK, Gugnani N, Gupta M. Efficacy of Different Precooling Agents and Topical Anesthetics on the Pain Perception during Intraoral Injection: A Comparative Clinical Study. Int J Clin Pediatr Dent. 2015 May-Aug;8(2):119-22. doi: 10.5005/jp-journals-10005-1296. Epub 2015 Aug 11. PMID 26379379
- [Background] Jayasuriya NSS, Weerapperuma ID, Amarasinghe MGCK. The use of an iced cotton bud as an effective pre-cooling method for palatal anaesthesia: A technical note. Singapore Dent J. 2017 Dec;38:17-19. doi: 10.1016/j.sdj.2017.07.001. PMID 29229069
- [Background] Bose S, Garg N, Pathivada L, Yeluri R. Cooling the soft tissue and its effect on perception of pain during infiltration and block anesthesia in children undergoing dental procedures: A comparative study. J Dent Res Dent Clin Dent Prospects. 2019 Summer;13(3):159-165. doi: 10.15171/joddd.2019.025. Epub 2019 Oct 7. PMID 31857860
- [Background] Tirupathi SP, Rajasekhar S. Effect of precooling on pain during local anesthesia administration in children: a systematic review. J Dent Anesth Pain Med. 2020 Jun;20(3):119-127. doi: 10.17245/jdapm.2020.20.3.119. Epub 2020 Jun 24. PMID 32617406
- [Background] Malanga GA, Yan N, Stark J. Mechanisms and efficacy of heat and cold therapies for musculoskeletal injury. Postgrad Med. 2015 Jan;127(1):57-65. doi: 10.1080/00325481.2015.992719. Epub 2014 Dec 15. PMID 25526231
- [Background] van Wijk AJ, Hoogstraten J. Anxiety and pain during dental injections. J Dent. 2009 Sep;37(9):700-4. doi: 10.1016/j.jdent.2009.05.023. Epub 2009 May 27. PMID 19556053
- [Background] Harbert H. Topical ice: a precursor to palatal injections. J Endod. 1989 Jan;15(1):27-8. doi: 10.1016/S0099-2399(89)80094-9. PMID 2607263
- [Background] Covino BG. Pharmacology of local anaesthetic agents. Br J Anaesth. 1986 Jul;58(7):701-16. doi: 10.1093/bja/58.7.701. PMID 2425835
- [Background] de Freiras GC, Pozzobon RT, Blaya DS, Moreira CH. Efficacy of Benzocaine 20% Topical Anesthetic Compared to Placebo Prior to Administration of Local Anesthesia in the Oral Cavity: A Randomized Controlled Trial. Anesth Prog. 2015 Summer;62(2):46-50. doi: 10.2344/0003-3006-62.2.46. PMID 26061572
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Sirintawat N, Sawang K, Chaiyasamut T, Wongsirichat N. Pain measurement in oral and maxillofacial surgery. J Dent Anesth Pain Med. 2017 Dec;17(4):253-263. doi: 10.17245/jdapm.2017.17.4.253. Epub 2017 Dec 28. PMID 29349347
- [Background] Hameed NN, Sargod SS, Bhat SS, Hegde SK, Bava MM. Effectiveness of precooling the injection site using tetrafluorethane on pain perception in children. J Indian Soc Pedod Prev Dent. 2018 Jul-Sep;36(3):296-300. doi: 10.4103/JISPPD.JISPPD_222_17. PMID 30246753
- [Background] Agrawal S, Sharma A, Dhurat R, Chahal K. The use of surgical gloves as an aseptic, effective, and inexpensive method to deliver circumferential cryoanesthesia. J Am Acad Dermatol. 2020 Jun;82(6):e195-e196. doi: 10.1016/j.jaad.2019.03.033. Epub 2019 Mar 21. No abstract available. PMID 30905796
- [Background] Ghaderi F, Banakar S, Rostami S. Effect of pre-cooling injection site on pain perception in pediatric dentistry: "A randomized clinical trial". Dent Res J (Isfahan). 2013 Nov;10(6):790-4. PMID 24379869
- [Background] Vafaei A, Rahbar M, Dadkhah R, Ranjkesh B, Erfanparast L. Children's Pain Perception and Behavioral Feedback during Local Anesthetic Injection with Four Injection Site Preparation Methods. Maedica (Bucur). 2019 Dec;14(4):343-349. doi: 10.26574/maedica.2019.14.4.343. PMID 32153664
- [Background] Pancekauskaite G, Jankauskaite L. Paediatric Pain Medicine: Pain Differences, Recognition and Coping Acute Procedural Pain in Paediatric Emergency Room. Medicina (Kaunas). 2018 Nov 27;54(6):94. doi: 10.3390/medicina54060094. PMID 30486427
- [Background] Flanagan T, Wahl MJ, Schmitt MM, Wahl JA. Size doesn't matter: needle gauge and injection pain. Gen Dent. 2007 May-Jun;55(3):216-7. PMID 17511363
- [Background] Dao TT, LeResche L. Gender differences in pain. J Orofac Pain. 2000 Summer;14(3):169-84; discussion 184-95. PMID 11203754
- [Background] Bagesund M, Tabrizi P. Lidocaine 20% patch vs lidocaine 5% gel for topical anaesthesia of oral mucosa. Int J Paediatr Dent. 2008 Nov;18(6):452-60. doi: 10.1111/j.1365-263X.2007.00910.x. Epub 2008 Mar 12. PMID 18341564
- [Background] Udeh C, Bittikofer J, Sum-Ping ST. Severe methemoglobinemia on reexposure to benzocaine. J Clin Anesth. 2001 Mar;13(2):128-30. doi: 10.1016/s0952-8180(01)00222-7. PMID 11331174
- [Background] Gonzalez-Rodriguez AJ, Gutierrez-Paredes EM, Revert Fernandez A, Jorda-Cuevas E. Allergic contact dermatitis to benzocaine: the importance of concomitant positive patch test results. Actas Dermosifiliogr. 2013 Mar;104(2):156-8. doi: 10.1016/j.ad.2011.07.023. Epub 2012 Apr 30. English, Spanish. PMID 22551703
- [Result] AmruthaVarshini I, Vinay C, Uloopi KS, RojaRamya KS, Chandrasekhar R, Penmatsa C. Effectiveness of Pre-cooling the Injection Site, Laser Biostimulation, and Topical Local Anesthetic Gel in Reduction of Local Anesthesia Injection Pain in Children. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):81-83. doi: 10.5005/jp-journals-10005-1913. PMID 34326589
- [Result] Wiswall AT, Bowles WR, Lunos S, McClanahan SB, Harris S. Palatal anesthesia: comparison of four techniques for decreasing injection discomfort. Northwest Dent. 2014 Jul-Aug;93(4):25-9. PMID 25233569
- [Result] Anantharaj A, Sabu JM, Ramakrishna S, Jagdeesh RB, Praveen P, Shankarappa PR. A comparative evaluation of pain perception following topical application of benzocaine gel, clove-papaya based anesthetic gel and precooling of the injection site before intraoral injections in children. J Indian Soc Pedod Prev Dent. 2020 Apr-Jun;38(2):184-189. doi: 10.4103/JISPPD.JISPPD_153_18. PMID 32611866
- See also: Related Info — https://www.iasp-pain.org/resources/terminology/
- See also: Related Info — https://www.wjoud.com/doi/pdf/10.5005/jp-journals-10015-1273
- See also: Related Info — https://jmcrr.info/index.php/jmcrr/article/view/44
- See also: Related Info — https://www.scielo.br/j/pboci/a/LRwW9FLLyNrNGQDgf6mWQnt/abstract/?lang=en